CLINICAL TRIAL: NCT01364519
Title: A Randomized, Double-Blind (3rd Party Open), Placebo-Controlled, 2-Way Crossover Study To Determine The Effects Of A Single Inhaled Dose Of 500 MCG Fluticasone Propionate On Induced Sputum Neutrophils Following Inhaled Lipopolysaccharide (LPS) Challenge In Healthy Volunteers
Brief Title: A Study To Determine Effects Of Fluticasone Propionate On Sputum Neutrophils After Inhaled Lipopolysaccharide Challenge In Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: A9011082
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Fluticasone Propionate
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo for Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Dry powder for inhalation, Single Dose, 500mcg
  Arms: Arm 1
Drug: Placebo for Fluticasone Propionate — Dry powder for inhalation, Single Dose, placebo
  Arms: Arm 2

SUMMARY:
Study to assess effect of Fluticasone Propionate on acute lung inflammation following inhaled lipopolysaccharide (LPS) challenge. Study will be conducted in healthy volunteers. Assessment of inflammation will be via sputum induction.

DETAILED DESCRIPTION:
Methodology Validation

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Normoresponsive airways - histamine PC20>16mg/mL
* Able to complete sputum induction successfully

Exclusion Criteria:

* Non (or ex) smokers
* No LPS challenge in previous 4 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Sputum Neutrophil (%) | 6 hours post LPS challenge

SECONDARY OUTCOMES:
Sputum Inflammatory cytokines (IL-6, MCP-1 and MIP1beta) | 6 hours post LPS challenge
Blood Inflammatory Cytokines (IL-6, MCP-1, fibrinogen, CC16, CRP and MIP1beta) | 1, 4 and 6 hours post LPS challenge
Sputum cells (macrophages and total cell count) | 6 hours post LPS challenge

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United Kingdom (2):
  - Pfizer Investigational Site, Manchester, Greater Manchester
  - Pfizer Investigational Site, London

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9011082&StudyName=A%20Study%20To%20Determine%20Effects%20Of%20Fluticasone%20Propionate%20On%20Sputum%20Neutrophils%20After%20Inhaled%20Lipopolysaccharide%20Challenge%20In%20Volunteers